CLINICAL TRIAL: NCT05888532
Title: A First-in-Human, Phase I/II PET Imaging Study of 64Cu-GRIP B, a Radiotracer Targeting Granzyme B, in Patients With Advanced Malignancies
Brief Title: 64Cu-GRIP B in Patients With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rahul Aggarwal (Other)
Collaborators: National Cancer Institute (NCI) (NIH); U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Rahul Aggarwal, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23921; NCI-2023-04001 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 5R01CA229354 (NIH); 5R01CA258297 (NIH)
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer; Renal Cancer; Urethral Cancer; Advanced Solid Tumor; Metastatic Castration-resistant Prostate Cancer; Solid Tumor, Adult
Keywords: Imaging Study; Radiotracer; Granzyme B
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms; Urethral Neoplasms; Lipodystrophy, Congenital Generalized | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: 64Cu-GRIP B, Solid Tumor Malignancy participants (Experimental): Participants with solid tumor malignancies (3 males, 3 females), dosimetry calculation will be performed by obtaining whole body (vertex to thighs) PET images up to five time points from 0.5 to 24 hours post 64Cu-GRIP B injections. An additional intravenous line will be placed in the contra-lateral arm to collect blood for this group.
  Interventions: Drug: Copper-64 labeled Granzyme B (64Cu-GRIP B); Procedure: Positron Emission Tomography (PET)
- Cohort B: 64Cu-GRIP B, RCC and UC participants (Experimental): Participants with renal cell and urothelial carcinoma will have longitudinal imaging performed prior to treatment outside of this study with anti-programmed death-1 (PD-1)/anti-PD-1 ligand 1 (PD-L1) blockade (with or without concomitant anti-CTLA4 treatment), after 8 weeks of checkpoint blockade, and again at the time of disease progression by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
  Interventions: Drug: Copper-64 labeled Granzyme B (64Cu-GRIP B); Procedure: Positron Emission Tomography (PET)
- Cohort C: 64Cu-GRIP B, mCRPC participants (Experimental): Participants with metastatic castration resistant prostate cancer (mCRPC)) will have longitudinal imaging performed prior to treatment outside of this study, 8 weeks following initiation of treatment outside of this study, and at the time of disease progression by Prostate Cancer Working Group 3 (PCWG3) criteria.
  Interventions: Drug: Copper-64 labeled Granzyme B (64Cu-GRIP B); Procedure: Positron Emission Tomography (PET)
- Cohort D: 64Cu-GRIP B, Advanced malignancies (Experimental): participants with solid tumor malignancies will have longitudinal imaging performed prior to treatment outside of this study, 8 weeks following initiation of treatment, and the opportunity to have an optional scan at the time of progression.
  Interventions: Drug: Copper-64 labeled Granzyme B (64Cu-GRIP B); Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: Copper-64 labeled Granzyme B (64Cu-GRIP B) — Given IV prior to imaging
  Other Names: 64Cu-GRIP B; 64Cu-labeled GRIP B
Procedure: Positron Emission Tomography (PET) — Imaging procedure
  Other Names: Positron Emission Tomography; PET; PET Scan

SUMMARY:
This phase I/II clinical trial evaluates if using a radiotracer targeting granzyme B, 64-copper granzyme targeting restricted interaction peptide specific to family member B (64 Cu-GRIP B) with positron emission tomography (PET) imaging can be safe and useful for detecting granzyme B (GrB) in patients with advanced cancers that has spread to nearby tissue or lymph nodes (advanced). Granzyme B (GrB) is a biomarker produced by immune cells in response to immunotherapy, which may highlight tumors that are more likely to respond to treatment. The study population is focused on genitourinary (GU) malignancies, including renal cell and urothelial cancer, two tumor types with high mutational burden and tumor infiltrating lymphocytes compared to other tumor types, and have a predictable response rate at the population level to immune checkpoint inhibitors. The information gained from this trial may allow researchers to develop future trials where 64Cu-GRIP B PET may serve as a biomarker to monitor early response to immunomodulatory therapies which are used to stimulate or suppress the immune system and may help the body fight cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, dosimetry, and pharmacokinetics of 64Cu-GRIP B PET in patients with solid tumor malignancy (3 males, 3 females). (Cohort A) II. To determine the mean percent change in both tumor maximum standardized uptake value (SUVmax) and ratio of SUVmax//blood average standardized uptake value (SUVave) on 64Cu-GRIP B PET in patients with participants with metastatic renal cell carcinoma (RCC) and urothelial carcinoma (UC) (Cohort B) or metastatic castration-resistant prostate cancer (mCRPC) (Cohort C).

SECONDARY OBJECTIVES:

I. To determine the safety and average organ dosimetry of 64Cu-GRIP B PET in patients with participants with metastatic RCC and UC (Cohort B), mCRPC (Cohort C) or other solid tumor malignancies (Cohort D).

II. To descriptively report the patterns of intra-tumoral uptake of 64Cu-GRIP B on whole body PET, including by site of disease, uptake by tumor type, inter-tumoral and inter-patient heterogeneity, and tumor-to-background signal in patients with participants with metastatic RCC and UC (Cohort B), mCRPC (Cohort C), or other solid tumor malignancies (Cohort D).

III. To descriptively report PET at grade >= 2 immune-related adverse event(s) in patients with metastatic RCC and UC (Cohort B) who have 64Cu-GRIP B PET performed within 14 days of onset of event.

IV. To descriptively report the number of lesions identified on 64Cu-GRIP B PET compared with conventional imaging in patients with participants with metastatic RCC and UC (Cohort B), mCRPC (Cohort C), or other solid tumor malignancies (Cohort D).

V. To determine whether baseline uptake on 64Cu-GRIP B PET is associated with subsequent clinical outcomes including objective response, progression-free survival, prostate-specific antigen 50% reduction (PSA50) response, and immune-related adverse events in participants with metastatic RCC and UC (Cohort B), mCRPC (Cohort C), or other solid tumor malignancies (Cohort D).

OUTLINE: Patients are assigned to 1 of 4 cohorts:

Cohort A: Participants with metastatic GU malignancy (renal,urothelial, or prostate) Cohort B: Participants with metastatic renal cell carcinoma (RCC) or urothelial cancer (UC).

Cohort C: Participants with mCRPC Cohort D: Participants with solid tumor malignancies

All participants will receive 64Cu-GRIP B PET at baseline. For participants in Cohorts B and C, another PET scan will be performed 8 weeks and at disease progression. Participants in Cohort D will undergo PET/CT or PET/MRI throughout the study and may undergo an optional 64Cu-GRIP B PET at the time of progression. Safety monitoring includes adverse event assessment at screening, 60 minutes (+/- 15 min), 2 hours (+/- 30 min), and 24 hours (+/- 4 hours) following 64Cu-GRIP B injections. Participants will be followed for up to 2 years for longitudinal endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Disease characteristics by cohort, as defined by:

   Cohort A:
   * Histologically-confirmed metastatic solid tumor malignancy (3 Male, 3 Female)
   * Locally advanced or metastatic disease on conventional imaging

   Cohort B:
   * Histologically-confirmed metastatic renal cell carcinoma (any histologic sub-type) or urothelial carcinoma
   * Locally advanced or metastatic disease on conventional imaging

   Cohort C:
   * Histologically-confirmed prostate adenocarcinoma
   * Metastatic castration resistant prostate cancer by Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria
2. Planned treatment with immune checkpoint inhibitor (Cohorts B and C only)
3. Willing to undergo paired tumor biopsies and has safely accessible bone or soft tissue lesion (Cohorts B and C only)
4. The subject is able and willing to comply with study procedures and provide signed and dated informed consent.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. Age 18 years or older at the time of study entry.
7. Adequate organ function, as defined by:

   * Serum creatinine <= 1.5 x upper limit of normal (ULN) or estimated creatinine clearance > 60 mL/min
   * Total bilirubin <= 1.5 x ULN (< 3 x ULN in patients with documented or suspected Gilbert's).
   * Hemoglobin >= 8.0 g/dL
   * Platelet count >= 75,000/microliter
   * Absolute neutrophil count ≥ 1000/microliter
8. Patients must not be pregnant or breast feeding. Women of childbearing potential are required to obtain a negative pregnancy test within 14 days of PET Imaging scan. Effective contraception (men and women) must be used in subjects of child-bearing potential.

Exclusion Criteria:

1. Patients who because of age, general medical or psychiatric condition, or physiologic status cannot give valid informed consent.
2. Any condition that, in the opinion of the Principal Investigator, would impair the patient's ability to comply with study procedures.
3. Is currently pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events (Cohort A) | Up to 8 weeks
  For Cohort A, the frequency and severity of adverse events following 64Cu-GRIP B injection will be descriptively reported, using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Percent of injected activity (Cohort A) | Up to 8 weeks
  For Cohort A, the tracer kinetics is measured in the organs and total-body, and the % of injected activity for each time point will be recorded for participants in Cohort A. This information is used as input for organ and whole-body effective dose calculation using Organ Level INternal Dose Assessment/EXponential Modeling (OLINDA/EXM). This will provide the data of whole-body effective dose (millisievert (mSv)/megabecquerels (MBq)), and organ doses.
Time to maximum observed concentration (Tmax) (Cohort A) | Up to 8 weeks
  Pharmacokinetic (PK) parameters for participants in Cohort A derived from plasma will be calculated using a non-compartmental approach with a log-linear terminal assumption for up to a possible 5 time points. A custom software package or a commercial software package like Phoenix WinNonlin will be used to compute the time it takes for a drug to reach the maximum concentration (Cmax) after administration of a drug that needs to be absorbed.
Maximum observed concentration (Cmax) (Cohort A) | Up to 8 weeks
  PK parameters for participants in Cohort A derived from plasma will be calculated using a non-compartmental approach with a log-linear terminal assumption for up to a possible 5 time points. A custom software package or a commercial software package like Phoenix WinNonlin will be used to compute the maximum concentration (Cmax) after administration of a drug that needs to be absorbed.
Area under the concentration-time curve (AUC) (Cohort A) | Up to 8 weeks
  PK parameters for participants in Cohort A derived from plasma will be calculated using a non-compartmental approach with a log-linear terminal assumption for up to a possible 5 time points. A custom software package or a commercial software package like Phoenix WinNonlin will be used to compute the area under the concentration-time curve (AUC) from hour 0 to the last measurable concentration (AUC0-t; min*unit/mL)
AUC extrapolated to infinity (Cohort A) | Up to 8 weeks
  PK parameters for participants in Cohort A derived from plasma will be calculated using a non-compartmental approach with a log-linear terminal assumption for up to a possible 5 time points. A custom software package or a commercial software package like Phoenix WinNonlin will be used to compute the AUC extrapolated to infinity (AUC0-∞; min*unit/mL)
Median clearance (Cohort A) | Up to 8 weeks
  PK parameters for participants in Cohort A derived from plasma will be calculated using a non-compartmental approach with a log-linear terminal assumption for up to a possible 5 time points. A custom software package or a commercial software package like Phoenix WinNonlin will be used to compute the volume of plasma which is completely cleared of a substance per minute (mL/min).
Apparent terminal elimination rate constant (Cohort A) | Up to 8 weeks
  PK parameters for participants in Cohort A derived from plasma will be calculated using a non-compartmental approach with a log-linear terminal assumption for up to a possible 5 time points. A custom software package or a commercial software package like Phoenix WinNonlin will be used to compute the apparent terminal elimination rate constant.
Apparent terminal elimination half-life (Cohort A) | Up to 8 weeks
  PK parameters for participants in Cohort A derived from plasma will be calculated using a non-compartmental approach with a log-linear terminal assumption for up to a possible 5 time points. A custom software package or a commercial software package like Phoenix WinNonlin will be used to compute apparent terminal elimination half-life (t1/2; min).
Change in SUVmax (Cohorts B, C, and D) | Up to 8 weeks
  For Cohorts B, C and D, descriptive statistics will be used to summarize the change in SUVmax from baseline to 8 weeks at lesion level for participants in Cohorts B & C.
Change in SUVmax/SUVave (Cohorts B, C, and D) | Up to 8 weeks
  For Cohorts B, C and D, descriptive statistics will be used to summarize the change in the ratio of SUVmax/SUVave from baseline to 8 weeks at lesion level for participants in Cohorts B & C.

SECONDARY OUTCOMES:
Frequency of treatment-emergent adverse events (Cohorts B, C, and D) | Up to 8 weeks
  For Cohorts B, C and D, the frequency and severity of adverse events following 64Cu-GRIP B injection will be descriptively reported
Mean SUVmax in metastatic lesions by disease site (Cohorts B, C and D) | Up to 2 years
  For Cohorts B, C and D, the mead/standard deviation (sd) (median and range, if normality assumption does not hold) for intra-tumoral SUVmax within metastatic lesions will be descriptively reported, to assess for intra-tumoral heterogeneity and differences in uptake by site of disease.
Percent of lesions detected for metastatic participants (Cohorts B, C and D) | Up to 8 weeks
  For Cohorts B, C and D, the percentage of metastatic lesions detected on conventional imaging that are also detected on baseline 64Cu-GRIP B PET will be descriptively reported with 95% confidence intervals.
Median change in SUVmax from baseline with reported immune-related adverse event (Cohort B) | Up to 2 years
  For the subset of patients in Cohort B experiencing Grade ≥ 2 immune-related adverse event who have 64Cu-GRIP B PET performed within 14 days of onset of event, the mean change from baseline in involved organ site(s) uptake on PET will be descriptively reported along with sd (or median with range) at lesion-level
Median change in SUVmax-ave from baseline with reported immune-related adverse event (Cohorts B) | Up to 2 years
  For the subset of patients in Cohort B experiencing Grade >= 2 immune-related adverse event who have 64Cu-GRIP B PET performed within 14 days of onset of event, the mean change from baseline in involved organ site(s) uptake on PET will be descriptively reported along with sd (or median with range) at patient-level
Association of baseline uptake with object response (ORR) (Cohorts B, C and D) | Up to 2 years
  For Cohort B, C and D , to analyze the association between the baseline in SUVmax and with subsequent response by RECIST 1.1 for Cohort B and modified RECIST 1.1/PCWG3 criteria, metastatic lesions will be segregated based on objective response by RECIST 1.1 criteria on follow up conventional imaging.
Association of baseline uptake with progression-free survival (PFS) (Cohorts B, C and D) | Up to 2 years
  For Cohorts B, C and D, to assess the association between the baseline SUVmax with progression-free survival, defined as the time from date of initiation of checkpoint inhibition to subsequent progression by Prostate Cancer Clinical Trials Working Group 3 (PCWG3)/RECIST criteria, the participant cohort will be dichotomized above and below the median PFS.
Association of baseline uptake with reported PSA50 response (Cohort C) | Up to 2 years
  For cohort C, to assess the association between the baseline in SUVmax with the patient cohort will be dichotomized into PSA50 vs. non-PSA50 responders.
Association of baseline uptake with reported immune-related adverse events (irAEs)(Cohorts B, C and D) | Up to 2 years
  For Cohorts B, C and D,to assess the association between the baseline in SUVmax with the patient cohort will be dichotomized into irAE vs. non-irAE reporters.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No